CLINICAL TRIAL: NCT01168739
Title: Effect of Combined Exercise, Heat, and Quercetin Supplementation on Whole Body Stress Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Gatorade Sports and Science Institute (Other); Quercegen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HRRC08-606
Record Dates: First submitted 2010-07-20; First posted 2010-07-23 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Heat Acclimation and Thermotolerance
Keywords: thermotolerance; heat acclimation; quercetin; exertional heat illness; gastrointestinal barrier permeability
MeSH Terms: conditions — Heat Stress Disorders | interventions — Quercetin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quercetin (Experimental): not necessary, contained in protocol
  Interventions: Dietary Supplement: Quercetin
- Placebo (Placebo Comparator): not necessary, contained in protocol
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Quercetin — 2g/d dietary quercetin supplementation, 1g taken am; 1g taken pm
  Arms: Quercetin
Dietary Supplement: Placebo — Placebo, performed on same subjects as Quercetin Arm, used to compare results between conditions
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether dietary quercetin supplementation effects thermotolerance and heat acclimation in human subjects exposed to exercise/heat stress.

Specific Aim I. To determine if quercetin in combination with repeated bouts of thermally stressful exercise will impact intestinal barrier function. The investigators will examine urinary lactulose excretion, plasma endotoxin,plasma quercetin, inflammatory cytokines (TNF-a & Il-6), anti-inflammatory cytokines (Il-10), and HSP70 and HSF-1 content of peripheral blood mononuclear cells.

Specific Aim II. To determine whether quercetin's suppresses the ability of human subjects to acclimate to exercise/heat stress. The investigators will examine body temperatures, heart rates, physiological strain, sweat and plasma volume responses to standardized heat tolerance tests.

DETAILED DESCRIPTION:
Overall Protocol:

This study will involve a repeated-measures design (2 conditions) in which subjects will perform exercise in the heat. Each condition will begin with an Intestinal Permeability Measurement (IP1), where subjects will be admitted to the General Clinical Research Center (GCRC), drinking a test solution and collecting their urine for 8 hours to measure intestinal integrity prior to heat stress. This will be followed by a Heat Tolerance Trial (HT1: 50min exercise at 50% VO2max in environmental chamber controlled at 56oC, 20%RF), used as a baseline measurement of subject's capacity to work in the heat. Following HT1 each subject will perform 7 Days of Heat Acclimation (HA)exercise (controlled hyperthermia design, each subject will elevate core temperature >39oC in 50min during 50 minutes of exercise in environmental chamber controlled at 56oC, 20%RF; rest 10 min in environmental chamber; then perform another 50min of exercise at this elevated core temperature). On days 1 and 7 of HA subjects will follow exercise by performing additional Intestinal Permeability Measurements, providing pre (IP2) and post acclimation (IP3) measurements of intestinal permeability. Day 6 of HA will provide a posttest measurement of subjects' capacity to work in the heat, and will be synonymous with Heat Tolerance Trial 2 (HT2).

Subjects will take quercetin during the seven days of HA in one condition, and placebo in the other. At least 1 month must elapse before a subject will be allowed to repeat the opposite condition. The order will be balanced (half will take quercetin first, the other half placebo). This will be a double blinded study. Neither the investigators nor the subjects will know whether a HA involves quercetin or placebo.

Due to the possibility of outside factors causing variations in intestinal permeability over the course of the study, IP1 will always be used as a baseline condition, with IP2 and IP3 being scored relative (as percent change) to the first. Subjects will never be supplemented in IP1, as this might affect basal measurements of permeability. However, because quercetin supplementation may only exert a transient effect on intestinal permeability, subjects will always be supplemented (with either placebo or quercetin, according to condition) in IP2 and IP3.

In all conditions, subjects will be required to follow guidelines on diet and exercise. They will be instructed to avoid caffeine, alcohol, and to stay well hydrated. They will be instructed to avoid exercise that is not directly outlined by the experiment (see attached). Their meals will be provided by the GCRC to ensure adequate nutrition and to avoid high dietary levels of quercetin. We are currently working with BioNutrition on this menu. To ensure compliance with this diet, subjects will fill out a food diary.

ELIGIBILITY:
Inclusion Criteria:

* Healthy: 1 or less CV risk factor. Positive risk factors include:

  * Family history
  * Current cigarette smoker or quit within the previous 6 months
  * Hypertension (>140/90 mmHg) or on antihypertensive medication
  * Impaired fasting glucose (>110 mg/dl)
  * Dyslipidemia (LDL>130 mg/dl;HDL<40 mg/dl, total >200 mg/dl)
  * Low VO2 peak: <40ml/kg/min
  * Overfatness(BMI>30 kg/m2 and/or body fat > 25%)
* Male
* 18-39 years of age
* Willing to follow study diet
* Willing to exercise for prescribed time
* Willing to tolerate hot environment
* Willing to avoid external influences (ambient heat, uv exposure, external exercise) for study duration

Exclusion Criteria:

* History of heat illness
* Current NSAID use
* Known gastrointestinal disease
* Illness (physician provide physical before subject begin each condition)

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Urinary Lactulose Excretion | Baseline
  Lactulose is a large molecule (disaccharide: 242 kDa) that should not be permeable to the gastrointestinal barrier under normal conditions.
  Subjects will ingest a test solution containing 10 g lactulose (Quintron Instrument Company, QT02500-10-5, Milwaukee, WI, USA) dissolved in 50 ml of distilled water. This is followed by 8 hour urine collection.
Plasma endotoxin | Baseline
  Plasma endotoxin will be detected with a standard limulus amebocyte lysate (LAL) kit (Cell Sciences, HIT302, Canton, MA, USA). The minimum and maximum detection limits of this kit are 1.4 pg/ml and 1,000 pg/ml, respectively.
Plasma Quercetin | Baseline
  Quercetin conjugates are hydrolysized from plasma with B-glucuronidase and arylsulfatase kit (Roche Diagnostics, 10127698001, Indianapolis, IN, USA). The resulting supernatant is applied to solid phase extraction cartridges and run through a vacuum manifold for purification. The eluent is 80% methanol / 20% 18 MOhm water. Following solid phase extraction chromatographic analysis is performed using high performance liquid chromatography (HPLC).
Plasma TNF-a | pre, post, 2hours post, 4 hours post exercise on Day 1 of exercise/heat stress
plasma Il-6 | Pre, post, 2hours post, 4 hours post exercise, day 1 of exercise/heat stress
Plasma Il-10 | Pre, post, 2 hours post, 4 hours post exercise on Day 1 of exercise/heat stress
HSP70 content of peripheral blood mononuclear cells | Pre, post, 2 hours post, 4 hours post exercise on day 1 of exercise/heat stress
HSF-1 content of peripheral blood mononuclear cells | Pre, post, 2 hours post, 4 hours post exercise on day 1 of exercise/heat stress
Core temperature response to heat tolerance test | heat tolerance test 1= before study onset
Skin temperature response to heat tolerance test | heat tolerance test 1= before study onset
Mean body temperature response to heat tolerance test | heat tolerance test 1= before study onset
Heart rate response to heat tolerance test | heat tolerance test 1= before study onset
Physiological strain response to heat tolerance test | heat tolerance test 1= before study onset
Urinary Lactulose Excretion | Day 1 of exercise/heat stress
Urinary Lactulose Excretion | Day 7 of exercise/heat stress
Plasma Quercetin | Day 1 of exercise/heat stress
Plasma Quercetin | Day 7 of exercise/heat stress
Plasma Endotoxin | Day 1 of exercise/heat stress
plasma endotoxin | day 7 of exercise/heat stress
Plasma TNF-a | pre, post, 2hours post, 4 hours post exercise on Day 7 of exercise/heat stress
plasma Il-10 | pre, post, 2hours post, 4 hours post exercise on Day 7 of exercise/heat stress
plasma Il-6 | pre, post, 2hours post, 4 hours post exercise on Day 7 of exercise/heat stress
HSP70 content of peripheral blood mononuclear cells | pre, post, 2hours post, 4 hours post exercise on Day 7 of exercise/heat stress
HSF-1 content of peripheral blood mononuclear cells | pre, post, 2hours post, 4 hours post exercise on Day 7 of exercise/heat stress
Core temperature response to heat tolerance test | heat tolerance trial 2 = day 6 of exercise/heat stress
Skin temperature response to heat tolerance test | heat tolerance trial 2 = day 6 of exercise/heat stress
Mean body temperature response to heat tolerance test | heat tolerance trial 2 = day 6 of exercise/heat stress
Heart rate response to heat tolerance test | heat tolerance trial 2 = day 6 of exercise/heat stress
physiological strain response to heat tolerance test | heat tolerance trial 2 = day 6 of exercise/heat stress

SECONDARY OUTCOMES:
Improvements in sweat rate following heat acclimation exercise | heat tolerance test 1= before study onset
Plasma volume expansion in response to heat acclimation exercise | heat tolerance test 1= before study onset
Improvements in sweat rate following heat acclimation exercise | heat tolerance trial 2 = day 6 of exercise/heat stress
plasma volume expansion in response to heat acclimation exercise | heat tolerance trial 2 = day 6 of exercise/heat stress

CONTACTS AND LOCATIONS:
Overall Officials: Pope L Moseley, MD, Principal Investigator — University of New Mexico, Professor and Chariman, Dpt of Internal Medicine; Matthew R. Kuennen, PhD, Study Director — UNM Department of Health, Exercise and Sports Sciences and UNM Department of Internal Medicine
Locations (1):
- UNM General Clinical Research Center, Albuquerque, New Mexico, United States